CLINICAL TRIAL: NCT02789696
Title: Prevalence of Acromegaly in a Diagnostic Consultation for Sleep Apnea Syndrome: A Prospective, National and Multicentric Study
Brief Title: Prevalence of Acromegaly in a Diagnostic Consultation for Sleep Apnea Syndrome
Acronym: ACROSAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13CHUG37
Record Dates: First submitted 2016-05-11; First posted 2016-06-03 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acromegaly (Other): Diagnosis of acromegaly
  Interventions: Other: Diagnosis of acromegaly

INTERVENTIONS:
Other: Diagnosis of acromegaly — Biological analysis of IGF-1

SUMMARY:
Prevalence of sleep apnea syndrome in patients with acromegaly is about 70%. It seems that comorbidities of arterial hypertension or type 2 diabetes are more severe in patients with acromegaly and sleep apnea syndrome. Besides sleep apnea syndrome associated to acromegaly gives rise to few symptoms, that explains it is under diagnosed. The mechanisms of the association are based on maxillofacial modifications linked to acromegaly, a thickening of soft tissues with deposits of glyco-aminoglycanes but probably also because of the associated obesity, of the potential existence of a goiter and a muscular dystrophy of the dilatative muscles of the pharynx.

At present, no study clearly documented prevalence of acromegaly in a diagnostic consultation for sleep apnea syndrome.

DETAILED DESCRIPTION:
60 investigators will participate to this study. They will be chosen among those participating to the sleep observatory of the federation of pneumology (www.osfp.fr).

All participating pneumologists would have to fill in the questionnaire (co-morbidities, concomitant treatments, biological analysis) directly online and also clinical signs and symptoms of acromegaly. A blood test for the insulin-like growth factor (IGF-1) dosage will be systematically prescribed to the patient. Pneumologists will have to include all consecutive patients presenting with sleep apnea syndrome suspicion.

According to first IGF-1 results, patients may have to do a second blood test in a referenced laboratory to confirm the dosage.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 40 kg/m2
* Patient consulting for sleep breathing disorder
* Informed consent signed
* patient covered by french health insurance

Exclusion Criteria:

* Other sleep disorder already diagnosed
* Pregnant women
* Patients participating in an other study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
determination of acromegaly prevalence | 1 year
  IGF-1 (insulin-like growth factor-1) quantification in blood punction

SECONDARY OUTCOMES:
description of clinical signs of acromegaly associated to sleep apnea syndrome (Epworth scale) | 1 year
  Score to Epworth scale will be compared between patients with sleep apnea syndrome with acromegaly and patients with sleep apnea syndrome only.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, Isère, France